CLINICAL TRIAL: NCT03717558
Title: Comparative Bioavailability Pilot Study of 3 W0035 Test Oral Suspensions (Ivermectin 1mg/mL) Versus Stromectol® (Ivermectin, 3 mg Tablet) After Single Oral Administration in Healthy Volunteers. Single Centre, Open Label, Crossover, Randomized, 5-period, 20-sequence, Partial Replicate, Single Dose Design
Brief Title: Bioavailability Pilot Study of Versus W0035 Versus Stromectol
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Pierre Fabre Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: W00035 PU 1 02
Record Dates: First submitted 2018-10-05; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Open label, crossover, randomized, 5-period, 20-sequence, partial replicate, single dose design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stromectol R (Active Comparator): Stromectol R = ivermectin 3mg (tablet)
  Interventions: Drug: ivermectin T1; Drug: ivermectin T2; Drug: ivermectin T3
- ivermectin T1 (Experimental): T1= ivermectin low grade particle Size Distribution
  Interventions: Drug: ivermectin T1; Drug: ivermectin T2; Drug: ivermectin T3
- ivermectin T2 (Experimental): T2= ivermectin medium grade particle Size Distribution
  Interventions: Drug: ivermectin T1; Drug: ivermectin T2; Drug: ivermectin T3
- ivermectin T3 (Experimental): T= ivermectin high grade particle Size Distribution
  Interventions: Drug: ivermectin T1; Drug: ivermectin T2; Drug: ivermectin T3

INTERVENTIONS:
Drug: ivermectin T1 — Subjects will be randomly assigned to one of the 20 different sequences of on single dose of ivermectin (T1, T2, and T3) and two single doses of Stromectol
Drug: ivermectin T2 — Subjects will be randomly assigned to one of the 20 different sequences of on single dose of ivermectin (T1, T2, and T3) and two single doses of Stromectol
Drug: ivermectin T3 — Subjects will be randomly assigned to one of the 20 different sequences of on single dose of ivermectin (T1, T2, and T3) and two single doses of Stromectol

SUMMARY:
Ivermectin is prescribed for the treatment of helminthic infections sensitive to ivermectin. However, it is currently only available as a tablet formulation. W0035 is a powder for oral suspension of ivermectin developed by PIERRE FABRE DERMATOLOGIE intended to be administered to children for the treatment of helminthic infections sensitive to ivermectin and mentioned in the Summary of Product Characteristics (SmPC) of Stromectol.

PIERRE FABRE DERMATOLOGIE intends to carry out this pilot bioavailability study in order to define the most appropriate formulation to be used in the bioequivalence study.

ELIGIBILITY:
Inclusion Criteria:

* 18.5 ≤ BMI ≤ 30.0 kg/m².
* Non-smoker subject with a breath carbon monoxide reading of ≤10 ppm at screening.
* Agree to use effective contraception method

Exclusion Criteria: most specific out of 30.

* History of or current symptomatic orthostatic hypotension
* Hyper-eosinophilia or subject at risk of microfilaremic disease or clinical suspicion of intestinal helminth infection
* History of or current macroscopic or microscopic hematuria
* Positive serology for Hepatitis Bs antigen (HBs), Hepatitis C Virus (HCV) and HIV 1 and 2 antibodies.
* Organic disorder likely to modify, absorption, distribution or elimination of the medication.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-30 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of ivermectin | 5 periods of 3 days each
  At each period: 17 blood samples: T0 (Pre-dose), T0 +15min, T0 +30min, T0 +1h, T0+1h30min, T0 +2h, T0 +2h30, T0 +3h, T0 +3h30, T0 +4h, T0 +4h30, T0 +5h, T0 +6h, T0 +12h, T0 +24h, T0 +48h and T0 +72h

CONTACTS AND LOCATIONS:
Overall Officials: Karim Keddad, MD, Study Director — Institut de Recherche Pierre Fabre
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No